CLINICAL TRIAL: NCT02061579
Title: Initiate and Maintain Physical Activity in Clinics: The IMPACT Diabetes Study
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Latha Palaniappan, MD, MS, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 31635; U.S. NIH Grant 5R18DK096394 (Other Grant/Funding Number: U.S. NIH Grant/Contract Award Number)
Record Dates: First submitted 2014-02-11; First posted 2014-02-13 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus
Keywords: Physical Activity
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Once-Weekly Structured Contact (Experimental): Participants in the Once Weekly Structured Contact group will take part in an 6-month exercise intervention and attend one structured group exercise session per week. They will engage in aerobic and resistance training for approximately 80 minutes per exercise session. Additionally, they will attend three exercise evaluations and six study visits.
  Interventions: Behavioral: Structured Group Exercise
- Thrice-Weekly Structured Contact (Experimental): Participants in the Thrice-Weekly Structured Contact group will take part in an 6-month exercise intervention and attend three structured group exercise sessions per week. In total, they will engage in aerobic and resistance training sessions for approximately 200 minutes per week. Additionally, they will attend three exercise evaluations and six study visits.
  Interventions: Behavioral: Structured Group Exercise
- Usual Care (No Intervention): Participants in the Usual Care group will not take part in an 6-month exercise intervention. They will continue to seek regular care from their primary care providers and attend six study visits.

INTERVENTIONS:
Behavioral: Structured Group Exercise — The study intervention is a 6-month exercise program with structured group sessions conducted in a clinical setting. Group sessions include Aerobic Training and Combined Training. Once-Weekly participants will attend one Combined Training session while thrice-weekly participants will attend two Combined Training sessions and one Aerobic Training session per week. Participants in both groups will attend three exercise evaluations during the intervention period. Participants will also use provided logs to track their daily exercise activities outside of group sessions. Physical activity will be assessed by group session attendance, exercise resistance and intensity, and exercise frequency data collected from exercise logs, surveys, and evaluations.
  Arms: Once-Weekly Structured Contact; Thrice-Weekly Structured Contact

SUMMARY:
The Initiate and Maintain Physical Activity in Clinics (IMPACT) study will determine the optimal and feasible level of frequency of structured contact needed in a clinical setting for adult patients with Type 2 Diabetes Mellitus to initiate and maintain physical activity recommendations long-term.

DETAILED DESCRIPTION:
The IMPACT Study will compare the health outcomes and lifestyle habits amongst the three groups of study participants. Study participants will be randomized into three exercise group. Group 1 will participate in instructor-led exercise training sessions 1 time per week, for 24 weeks (approximately 6 months). Group 2 will participate in instructor-led exercise training sessions 3 times per week, for 24 weeks (approximately 6 months). Group 3 will not attend any instructor-led exercise training sessions. All groups will be encouraged to see their usual providers for routine healthcare, and continue their usual medication regimen.

ELIGIBILITY:
Inclusion Criteria:

* Recent hemoglobin A1c result between 6.5 and 13.0%
* Diagnosed with Type 2 Diabetes Mellitus
* Able and willing to enroll and meet the requirements of the study

Exclusion Criteria:

* Inability to speak, read or understand English
* Long-term current use or dependency on insulin
* Systolic blood pressure >180 mm Hg or diastolic blood pressure >100 mm Hg
* Resting heart rate > 120 bpm
* History of or present heart or cardiovascular conditions
* History of or present respiratory disease
* History of or present spinal cord injury
* History of stroke or Transient Ischemic Attack (TIA)
* History of cancer diagnosis in the past 5 years or present cancer diagnosis
* Medical, psychiatric, behavioral limitations that may interfere with study participation
* Participating in other clinical trials that may interfere with study procedures and outcomes
* Currently pregnant or plans to become pregnant within three years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Changes in Hemoglobin A1c Level Across Study Visits | Baseline, 3-, 6-, 18-, 24-, 30-month follow-up
Changes in Maximal Oxygen Consumption Across Study Visits | Baseline, 3-, 6-, 18-, 24-, 30-month follow-up
Changes in Self-Reported Physical Activity Level Across Study Visits | Baseline, 3-, 6-, 18-, 24-, 30-month follow-up

SECONDARY OUTCOMES:
Changes in Body Weight Across Study Visits | Baseline, 3-, 6-, 18-, 24-, 30-month follow-up
Changes in Body Mass Index Across Study Visits | Baseline, 3-, 6-, 18-, 24-, 30-month follow-up
Changes in Waist Circumference Across Study Visits | Baseline, 3-, 6-, 18-, 24-, 30-month follow-up
Changes in Blood Pressure Across Study Visits | Baseline, 3-, 6-, 18-, 24-, 30-month follow-up
Changes in Heart Rate Across Study Visits | Baseline, 3-, 6-, 18-, 24-, 30-month follow-up
Changes in Dietary Intake Across Study Visits | Baseline, 3-, 6-, 18-, 24-, 30-month follow-up
Changes in Self-Reported Quality of Life Across Study Visits | Baseline, 3-, 6-, 18-, 24-, 30-month follow-up
Changes in Exercise Perception Across Study Visits | Baseline, 6-, 30-month follow-up
Changes in Patient Satisfaction During Intervention Period | 3-, 6-month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

REFERENCES:
- [Derived] Mukherji AB, Lu D, Qin F, Hedlin H, Johannsen NM, Chung S, Kobayashi Y, Haddad F, Lamendola C, Basina M, Talamoa R, Myers J, Palaniappan L. Effectiveness of a Community-Based Structured Physical Activity Program for Adults With Type 2 Diabetes: A Randomized Clinical Trial. JAMA Netw Open. 2022 Dec 1;5(12):e2247858. doi: 10.1001/jamanetworkopen.2022.47858. PMID 36542382